CLINICAL TRIAL: NCT04603248
Title: A Study for Identification of Immune Determinants for Response to Nivolumab in Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Chang Gon Kim, Principal Investigator, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4-2020-0801
Record Dates: First submitted 2020-10-08; First posted 2020-10-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: Head and Neck Squamous Cell Carcinoma (HNSCC)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 3mg/kg treatment will be given every 2 weeks up to progression or unacceptable toxicity

SUMMARY:
A study for identification of immune determinants for response to Nivolumab in Recurrent /Metastatic HNSCC(Head and neck squamous cell carcinoma) patients.

Recurrent and metastatic head and neck squamous cell carcinoma is incurable and requires aggressive treatment, resulting in functional disability, dismal prognosis, and high mortality rate. Prognosis of Recurrent and metastatic head and neck squamous cell carcinoma is poor, with limited treatment options and survival rates of 6-9 months following standard-of-care (SOC) therapies. Clinical trials have demonstrated promising clinical activity of anti PD-1(programmed death-1) therapy in head and neck squamous cell carcinoma. Currently, nivolumab were approved for head and neck squamous cell carcinoma refractory to platinum-based therapy. However, the response rate of anti PD-1(programmed death-1) therapy is relatively low and durable clinical benefit is limited to the minority of patients. Moreover, the presence of PD-1(programmed death-1) did not clearly predict response and treatment survival outcome, reflecting imperfection of this biomarker. Actually, PD-1(programmed death-1) negativity cannot preclude the therapeutic benefit of PD-1(programmed death-1) blockade, and vice versa. Hence, development of reliable predictive biomarkers is essential for proper patient selection to maximize clinical benefit of PD-1(programmed death-1) blockade in head and neck squamous cell carcinoma patients.

Therefore, we need to select patients who are most likely to benefit from anti PD-1(programmed death-1) therapy and identify the better biomarker to predict the response to PD-1(programmed death-1) blockade in head and neck squamous cell carcinoma patients. patients earlier than tumor assessment by imaging scan.

In the current study, we aimed to elucidate immune-related biomarkers to predict response with tumor tissue and peripheral blood from Recurrent /Metastatic HNSCC(Head and neck squamous cell carcinoma) patients treated with nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: Male or female
2. Age (at the time of informed consent): 19 years and older
3. Subjects with histologically- or cytologically-confirmed recurrent and/or metastatic head and neck squamous cell carcinoma (Recurrent/Metastatic HNSCC)
4. Known human papilloma virus (HPV) infection status with p16 immunohistochemistry or HPV in-situ hybridization
5. Failed or intolerable to previous platinum-based chemotherapy
6. Patients who have at least 1 measurable or non-measurable lesion per the RECIST (Response Evaluation Criteria in Solid Tumor) Guideline Ver. 1.1 as confirmed by imaging within 28 days before enrollment. The following requirements should also be satisfied:

   * If patients only have lesions that were previously treated with radiation, the lesion should be limited to one with confirmed aggravation by imaging after radiation.
   * If patients have pericardial or pleural effusion or ascites only, the lesion should be limited to one with cytologically confirmed malignancy.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
8. Patients with a life expectancy of at least 3 months
9. Screening laboratory values within the specified ranges stated below, obtained within 14 days prior to first dose:

   * White blood cells ≥2,000/mm3 and neutrophils ≥1,500/mm3
   * Platelets ≥100,000/mm3
   * Hemoglobin ≥9.0 g/dL
   * AST (GOT) and ALT (GPT) ≤3.0-fold the upper limit of normal (ULN) of the study site (or ≤5.0-fold the ULN of the study site in patients with liver metastases)
   * Total bilirubin ≤1.5-fold the ULN of the study site
   * Creatinine ≤1.5-fold the ULN of the study site or creatinine clearance (either the measured or estimated value using the Cockcroft-Gault equation) >45 mL/min
10. Explicit and voluntary consent to participate in the study obtained using a signed and dated informed consent form clearly and fully describing the purpose, potential risks, and any other critical issues regarding the study
11. Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons#1) must agree to use contraception(#2) from the time of informed consent until 5 months or more after the last dose of the investigational product. Also, women must agree not to breastfeed from the time of informed consent until 5 months or more after the last dose of the investigational product
12. Men must agree to use contraception(#2) from the start of study treatment until 7 months or more after the last dose of the investigational product.

    * #1 Women of childbearing potential are defined as all women after the onset of menstruation who are not postmenopausal and have not been surgically sterilized (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy). Postmenopause is defined as amenorrhea for ≥12 consecutive months without specific reasons. Women using oral contraceptives, intrauterine devices, or mechanical contraception such as contraceptive barriers are regarded as having childbearing potential.
    * #2 The subject must consent to use any two of the following methods of contraception: vasectomy or condom for patients who are male or female subject's partner and tubal ligation, contraceptive diaphragm, intrauterine device, spermicide, or oral contraceptive for patients who are female or male subject's partner.

Exclusion Criteria:

1. Patients with multiple primary cancers (with the exception of completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, or superficial bladder cancer, or any other cancer that has not recurred for at least 3 years)
2. Patients with residual adverse effects of prior therapy or effects of surgery that would affect the safety evaluation of the investigational product in the opinion of the investigator or sub-investigator.
3. Patients with current or past history of severe hypersensitivity to any other antibody products
4. Patients with concurrent autoimmune disease or history of chronic or recurrent autoimmune disease
5. Patients with a current or past history of interstitial lung disease or pulmonary fibrosis diagnosed based on imaging or clinical findings. Patients with radiation pneumonitis may be enrolled if the radiation pneumonitis has been confirmed as stable (beyond acute phase) without any concerns about recurrence.
6. Patients with concurrent diverticulitis or symptomatic gastrointestinal ulcerative disease
7. Patients with any metastasis in the brain or meninx that is symptomatic or requires treatment. Patients may be enrolled if the metastasis is asymptomatic and requires no treatment.
8. Patients with pericardial fluid, pleural effusion, or ascites requiring treatment
9. Patients with uncontrollable, tumor-related pain
10. Patients who have experienced medically refractory transient ischemic attack, cerebrovascular accident, thrombosis, or thromboembolism (pulmonary arterial embolism or deep vein thrombosis) within 180 days before enrollment
11. Patients with a history of uncontrollable or significant cardiovascular disease meeting any of the following criteria:

    * Myocardial infarction within 180 days before enrollment
    * Uncontrollable angina pectoris within 180 days before enrollment
    * New York Heart Association (NYHA) Class III or IV congestive heart failure
    * Uncontrollable hypertension despite appropriate treatment (e.g., systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥ 90 mmHg lasting 24 hours or more)
    * Arrhythmia requiring treatment
12. Patients with uncontrollable diabetes mellitus
13. Patients with systemic infections requiring treatment with intravenous antibiotics
14. Patients who have received systemic corticosteroids (more than 10mg/day prednisolone except for temporary use, e.g., for examination or prophylaxis of allergic reactions) or immunosuppressants within 28 days before enrollment
15. Patients who have received antineoplastic drugs (e.g., chemotherapy agents, molecular-targeted therapy agents, or immunotherapy agents) within 14 days before enrollment
16. Patients who have undergone surgical adhesion of the pleura or pericardium within 14 days before enrollment
17. Patients who have undergone surgery under general anesthesia within 14 days before enrollment
18. Patients who have undergone surgery involving local or topical anesthesia within 7 days before enrollment
19. Patients who have received radiotherapy within 14 days before enrollment, or radiotherapy to bone metastases within 7 days before enrollment
20. Patients who have received any radiopharmaceuticals (except for examination or diagnostic use of radiopharmaceuticals) within 56 days before enrollment
21. Patients with a positive test result for any of the following: HIV-1 antibody, HIV-2 antibody, HTLV-1 antibody, HBs antigen, or HCV antibody
22. Patients with a negative HBs antigen test but a positive test result for either HBs antibody or HBc antibody with a detectable level of HBV-DNA
23. Women who are pregnant or breastfeeding, or possibly pregnant
24. Patients who have received any other unapproved drug (e.g., investigational use of drugs, unapproved combined formulations, or unapproved dosage forms) within 28 days before enrollment
25. Patients who have previously received Nivolumab, anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, anti-CD137 antibody, anti-CTLA-4 antibody or other therapeutic antibodies or pharmacotherapies for regulation of T-cells
26. Patients judged to be incapable of providing consent for reasons such as concurrent dementia
27. Other patients judged by the investigator or sub-investigator to be inappropriate as subjects of this study
28. Patient with current or past history of hypersensitivity to Nivolumab.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Explore the biomarkers to predict objective response (OR) | Screening
  Single cell RNA sequencing (scRNA-seq), Multiplex IHC (Vectra Polaris®), T cell immunophenotyping using flow cytometry, papilloma virus (HPV) infection status with p16 immunohistochemistry or HPV in-situ hybridization, Microbiome, Evaluation of PD-L1 expression status based on combined positivity score and tumor rate score
Explore the biomarkers to predict objective response (OR) | Before Cycle2 Day1 (each cycle is 14 days)
  Single cell RNA sequencing (scRNA-seq), Multiplex IHC (Vectra Polaris®), T cell immunophenotyping using flow cytometry, papilloma virus (HPV) infection status with p16 immunohistochemistry or HPV in-situ hybridization, Evaluation of PD-L1 expression status based on combined positivity score and tumor rate score
Explore the biomarkers to predict objective response (OR) | From date of randomization until the date of first documented progression or date of unacceptable toxicity, whichever came first, assessed up to 100 months
  Single cell RNA sequencing (scRNA-seq), Multiplex IHC (Vectra Polaris®), T cell immunophenotyping using flow cytometry, papilloma virus (HPV) infection status with p16 immunohistochemistry or HPV in-situ hybridization, Evaluation of PD-L1 expression status based on combined positivity score and tumor rate score
Explore the biomarkers to predict progression-free survival (PFS) | Screening
  Single cell RNA sequencing (scRNA-seq), Multiplex IHC (Vectra Polaris®), T cell immunophenotyping using flow cytometry, papilloma virus (HPV) infection status with p16 immunohistochemistry or HPV in-situ hybridization, Microbiome, Evaluation of PD-L1 expression status based on combined positivity score and tumor rate score
Explore the biomarkers to predict progression-free survival (PFS) | Before Cycle2 Day1 (each cycle is 14 days)
  Single cell RNA sequencing (scRNA-seq), Multiplex IHC (Vectra Polaris®), T cell immunophenotyping using flow cytometry, papilloma virus (HPV) infection status with p16 immunohistochemistry or HPV in-situ hybridization, Evaluation of PD-L1 expression status based on combined positivity score and tumor rate score
Explore the biomarkers to predict progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of unacceptable toxicity, whichever came first, assessed up to 100 months
  Single cell RNA sequencing (scRNA-seq), Multiplex IHC (Vectra Polaris®), T cell immunophenotyping using flow cytometry, papilloma virus (HPV) infection status with p16 immunohistochemistry or HPV in-situ hybridization, Evaluation of PD-L1 expression status based on combined positivity score and tumor rate score
Explore the biomarkers to predict overall survival (OS) | Screening
  Single cell RNA sequencing (scRNA-seq), Multiplex IHC (Vectra Polaris®), T cell immunophenotyping using flow cytometry, papilloma virus (HPV) infection status with p16 immunohistochemistry or HPV in-situ hybridization, Microbiome, Evaluation of PD-L1 expression status based on combined positivity score and tumor rate score
Explore the biomarkers to predict overall survival (OS) | Before Cycle2 Day1 (each cycle is 14 days)
  Single cell RNA sequencing (scRNA-seq), Multiplex IHC (Vectra Polaris®), T cell immunophenotyping using flow cytometry, papilloma virus (HPV) infection status with p16 immunohistochemistry or HPV in-situ hybridization, Evaluation of PD-L1 expression status based on combined positivity score and tumor rate score
Explore the biomarkers to predict overall survival (OS) | From date of randomization until the date of first documented progression or date of unacceptable toxicity, whichever came first, assessed up to 100 months
  Single cell RNA sequencing (scRNA-seq), Multiplex IHC (Vectra Polaris®), T cell immunophenotyping using flow cytometry, papilloma virus (HPV) infection status with p16 immunohistochemistry or HPV in-situ hybridization, Evaluation of PD-L1 expression status based on combined positivity score and tumor rate score

SECONDARY OUTCOMES:
Safety: Number of participants with adverse events and abnormal laboratory values as assessed by NCI-CTCAE version 5 | From date of randomization until the date of first documented progression or date of unacceptable toxicity, whichever came first, assessed up to 100 months
  Number of participants with adverse events and abnormal laboratory values as assessed by NCI-CTCAE version 5

CONTACTS AND LOCATIONS:
Overall Officials: Hye Ryun Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided